CLINICAL TRIAL: NCT06840210
Title: Transforming Kidney Care in the Emergency Department: A Prospective Effectiveness-Implementation Evaluation
Brief Title: Effectiveness-Implementation Evaluation of Acute Kidney Injury Decision Support
Acronym: AKIDS
Status: Not yet recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Agency For Healthcare Research & Quality (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00367884; R01HS027793 (AHRQ)
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; AKI; Prediction; Machine Learning; Emergency Department; Clinical Decision Support
MeSH Terms: conditions — Acute Kidney Injury; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 365 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All adult ED patients with creatinine concentration measured during the participant's ED stay

SUMMARY:
Study Purpose: This study is testing an artificial intelligence (AI)-powered clinical decision support (CDS) system designed to help emergency department (ED) doctors detect and manage acute kidney injury (AKI) earlier. The goal is to see whether the tool improves patient care, clinician decision-making, and hospital outcomes when used in real-world ED settings.

Study Design:

The AI tool will be gradually introduced at three hospital EDs:

Johns Hopkins Hospital (JHH) Bayview Medical Center (BMC) Howard County General Hospital (HCGH)

Before the tool is activated, it will run in the background to collect baseline data without influencing care. Once implemented, doctors will receive training, and researchers will track how often the tool is used and whether it improves AKI care.

What the Study Measures:

Process Outcomes: Does the tool help doctors identify AKI sooner, avoid harmful medications, and improve decision-making about hospitalization?

Clinical Outcomes: Does the tool reduce the number and severity of AKI cases and improve kidney-related health outcomes?

Implementation Outcomes: Do ED doctors find the tool useful? Does it fit into the ED doctor's workflow without slowing the ED doctor's down?

Expected Impact: If successful, the AI tool could be expanded to other hospitals and used to improve early detection and treatment of AKI, reducing kidney complications and improving patient care nationwide.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following conditions to be eligible for the study:

1. Emergency Department Visit

   Patients presenting to one of the three study site emergency departments (EDs):

   Johns Hopkins Hospital (JHH) Bayview Medical Center (BMC) Howard County General Hospital (HCGH) Serum Creatinine Measurement
2. At least one serum creatinine (sCr) test performed during the ED visit.
3. Age: Adults (≥18 years old) at the time of ED visit.
4. Follow-Up Data Available: To be included in analysis for the investigator's secondary effectiveness outcome (new or progressive AKI) patients must have repeat creatinine concentration measurement available within 72 hours

Exclusion Criteria:

1. No ED Serum Creatinine Data: Patients who do not have a measured serum creatinine (sCr) value during the ED visit will not have decision support provided during the ED stay.
2. Patients Discharged Without Follow-Up Data: Patients discharged from the ED who do not undergo a follow-up serum creatinine test within 72 hours will be excluded from analysis of new or progressive AKI outcome assessment.
3. Age <18 Years
4. End-Stage Kidney Disease (ESKD) or Chronic Dialysis: Patients with a documented history of end-stage kidney disease (ESKD), (patients receiving chronic dialysis (hemodialysis or peritoneal dialysis) will will be excluded from analysis of new or progressive AKI outcome assessment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency Department
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Patients who receive Guideline-Concordant Kidney Care | From time of decision support provision until departure from the ED, approximately 6 hours

SECONDARY OUTCOMES:
New or Progressive Acute Kidney Injury | Within 72 hours of first creatinine measurement in the ED
Perceived usefulness and usability of AKIDS software as assessed by the System Usability Score | Prior to AKIDS implementation, immediately after implementation, and post implementation 6 months
  Will be assessed using the usability using the System Usability Score, a 10-item Likert scale that yields a single composite score on a scale of 0-100, with 100 being most usable.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremiah Hinson, MD, PhD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No